CLINICAL TRIAL: NCT00634348
Title: A Four-Week Double Blind Multicenter Study Comparing The Efficacy And Safety Of Ziprasidone To Aripiprazole In Subjects With Schizophrenia Or Schizoaffective Disorder Needing Inpatient Care
Brief Title: A Study Comparing the Efficacy and Safety of Ziprasidone and Aripiprazole for the Treatment fo Schizophrenia or Schizoaffective Disorder in Hospitalized Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1281110
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole; ziprasidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aripiprazole (Active Comparator)
  Interventions: Drug: Aripiprazole
- Ziprasidone (Active Comparator)
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Aripiprazole — Oral aripiprazole capsules 15 mg once daily from Days 1-14; thereafter, doses could be adjusted on Days 14 and 21 to 10, 15, or 30 mg once daily; patients treated for 28 days
  Arms: Aripiprazole
Drug: Ziprasidone — Oral ziprasidone capsules 40 mg twice daily on Day 1, 60 mg twice daily on Day 2, 80 mg twice daily on Days 3-14; thereafter, doses could be adjusted on Days 14 and 21 to 40, 60, or 80 mg twice daily; patients treated for 28 days
  Arms: Ziprasidone

SUMMARY:
The purpose of this study is to compare the efficacy and safety of ziprasidone and aripiprazole in hospitalized patients with schizophrenia or schizoaffective disorder

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with schizophrenia or schizoaffective disorder
* At least a 6th grade reading level
* Males or females, between 18 and 70 years of age at the time of consent
* Subjects must have been hospitalized for no more than 14 consecutive days immediately prior to screening

Exclusion Criteria:

* Psychiatric disorder other than schizophrenia or schizoaffective disorder
* History of arrhythmia, heart attack, or heart failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2004-04; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline to endpoint in Clinical Global Impressions-Severity (CGI-S) scale scores. | 28 days
Change from baseline to endpoint in Brief Psychiatric Rating Scale derived (BPRSd) total scores. | 28 days

SECONDARY OUTCOMES:
Change from baseline to Days 2, 4, 7, 14, 21, and 28 in Positive and Negative Syndrome Scale (PANSS) positive subscale scores. | 28 days
Change from baseline to Days 2, 4, 7, 14, 21, and 28 in PANSS negative subscale scores. | 28 days
Change from baseline to Days 2, 4, 7, 14, 21, and 28 in PANSS Depression factor scores. | 28 days
Change from baseline to endpoint in Calgary Depression Scale for Schizophrenia (CDSS) scores. | 28 days
Change from baseline to Days 2, 4, 7, 14, 21, and 28 in COVI Anxiety Scale scores. | 28 days
Change from baseline to endpoint in Global Assessment of Functioning (GAF) scale scores. | 28 days
Change from baseline to endpoint in Drug Attitude Inventory (DAI) scores. | 28 days
Change from baseline to endpoint in Personal Evaluation of Transition in Treatment (PETiT) scale scores. | 28 days
Change from baseline to endpoint in Patient Preference Scale (PPS) scores. | 28 days
Change from baseline to endpoint in Life Skills Profile (LSP). | 28 days
Change from baseline in Outcome Resource Discharge Questionnaire (ORDQ) scores on Days 2, 4, 7, 14, 21, and 28. | 28 days
Change from baseline to endpoint in Cognitive Battery. | 28 days
Change from baseline to Days 2, 4, 7, 14, 21, and 28 in PANSS total scores. | 28 days
Change from baseline to Days 2, 4, 7, 14, 21, and 28 in Clinical Global Impressions-Improvement (CGI-I) scale scores. | 28 days
Adverse events, laboratory evaluations, vital signs, electrocardiograms at baseline and on Days 2, 4, 7, 14, 21, and 28. | 28 days
Change from baseline to Day 28 in movement disorder rating scale scores. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- United States (36):
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Cerritos, California
  - Pfizer Investigational Site, Culver City, California
  - Pfizer Investigational Site, Garden Grove, California
  - Pfizer Investigational Site, Glendale, California
  - Pfizer Investigational Site, La Mesa, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Paramount, California
  - Pfizer Investigational Site, Riverside, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Hialeah, Florida
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Rockville, Maryland
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Clementon, New Jersey
  - Pfizer Investigational Site, Princeton, New Jersey
  - Pfizer Investigational Site, Willingboro, New Jersey
  - Pfizer Investigational Site, Woodlane, New Jersey
  - Pfizer Investigational Site, Jamaica, New York
  - Pfizer Investigational Site, Staten Island, New York
  - Pfizer Investigational Site, Butner, North Carolina
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Bellaire, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Irving, Texas
  - Pfizer Investigational Site, Arlington, Virginia
  - Pfizer Investigational Site, Falls Church, Virginia